CLINICAL TRIAL: NCT03862872
Title: The Effects of Oral Supplementation With Bend Beauty's Anti-Aging Formula on Inflammatory Markers
Brief Title: Effects of Bend Beauty's Anti-Aging Formula on Inflammatory Markers
Acronym: BENCHMARK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Altered research priorities
Sponsor: Bend Beauty Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT1801
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2019-12

CONDITIONS: Inflammation; Skin Abnormalities; Skin Pigment; Inflammatory Response; Skin Inflammation
Keywords: Inflammation; Skin; UV-light; Inflammatory markers; Eicosapentaenoic acid (EPA); Docosahexaenoic acid (DHA); Fish Oil; Gamma-linolenic acid (GLA); Borage oil; Vitamin D; Zeaxanthin; Lutein; Omega-3 Index; Chronic Inflammation Test; 11-dehydrothromboxane B2; 8-hydroxy-2' -deoxyguanosine (8- OHdG); 8-isoprostane
MeSH Terms: conditions — Inflammation; Skin Abnormalities; Pigmentation Disorders; Dermatitis

STUDY DESIGN:
Intervention Model Description: Phase IV, randomized, double-blind, placebo-controlled, three-arm, parallel intervention study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subject Code Numbers assigned to subjects using 400 randomly generated numbers ranging from 1-1000 are associated with all data generated in place of the subject name.
  Product Code Numbers on Test Materials, using 90 randomly generated numbers ranging from 1-99, are assigned by a Data Manager. All subsequent documentation will be labelled with the Product Code Number. Test material identity will not be shared with any participants within the trial [i.e. Subjects, Principal Investigator (PI), Clinical Research Monitor (CRM), Test Material Controller (TMC), Study Site Monitor & Quality Specialist (SM&QS), Data Analyst]. The only person who will be aware of the test material identity relative to any Product Code Number will be the Data Manager.
  Unmasking of the Product Code Numbers will be by the Data Manager, once statistical analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anti-Aging Formula (Experimental): 4 capsules daily of high-EPA fish oil, borage oil, zeaxanthin, lutein and vitamin D providing 1050 mg of Eicosapentaenoic acid (EPA) and 350 mg of Docosahexaenoic acid (DHA), 120 mg of Gamma-linolenic acid (GLA), 2.5 mg of zeaxanthin, 5 mg of lutein and 25 μg (1000 IU) of vitamin D3 for 90 days.
  Interventions: Dietary Supplement: Anti-Aging Formula
- Control Fish Oil (Active Comparator): 4 capsules daily of 1,106 mg each of triglyceride fish oil from anchovies, sardines, and/or mackerel whole body oil providing 816 mg EPA and 572 mg DHA total for 90 days.
  Interventions: Dietary Supplement: Control Fish Oil
- Inert Placebo (Placebo Comparator): 4 capsules daily of 1040 mg each of corn oil for 90 days.
  Interventions: Other: Inert Placebo

INTERVENTIONS:
Dietary Supplement: Anti-Aging Formula — Anti-Aging Formula contains 1050 mg of EPA and 350 mg of DHA from anchovies, sardines, and/or mackerel whole body oil, 120 mg of GLA from Borage (Borago officianalis) seeds, 2.5 mg of zeaxanthin from Capsicum annuum L. fruit, 5 mg of lutein from Tagetes erecta flower, and 25 μg (1000 IU) of vitamin D3 (cholecalciferol) from lanolin per 4 capsule daily dose. This dosage form is the same as is commercially marketed in Canada under license Natural Product Number (NPN) 80077254.
  Other Names: Bend Beauty's Anti-Aging Formula
  Arms: Anti-Aging Formula
Dietary Supplement: Control Fish Oil — The control fish oil is a soft gelatin capsule containing 1,106 mg of triglyceride fish oil from anchovies, sardines, and/or mackerel whole body oil. A four capsule per day dose provides 816 mg EPA and 572 mg DHA, which is only slightly less EPA+DHA than is provided within a four capsule per day dose of Anti-Aging Formula. This minor difference would not be expected to alter clinical outcomes.
  Arms: Control Fish Oil
Other: Inert Placebo — The inert placebo is a soft gelatin capsule containing 1040 mg of corn oil.
  Arms: Inert Placebo

SUMMARY:
This is a phase IV, randomized, double-blind, placebo-controlled, three-arm, parallel intervention study including three groups of 25 subjects between 35-65 years of age, treated with either Bend Beauty's Anti-Aging Formula, fish oil control or inert placebo for 90 days, with testing points at baseline, 30, 60, and 90 days.

DETAILED DESCRIPTION:
This is a phase IV, randomized, double-blind, placebo-controlled, three-arm, parallel intervention study including three groups of 25 subjects between 35-65 years of age, treated with either Bend Beauty's Anti-Aging Formula, fish oil control or inert placebo for 90 days, with testing points at baseline, 30, 60, and 90 days.

Subjects will be preselected through a Subject Eligibility Screening (SES) against defined inclusion and exclusion criteria for entry into the trial. Eligible participants will be tested using the Chronic Inflammation Test for urinary 11-dehydrothromboxane B2 (https://chronicinflammationtest.com) and the Omega-3 Index Test for eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) in red blood cells (RBC) (https://omegaquant.com ), to confirm possible presence of chronic inflammation. If these test results meet a defined limit, participants will be enrolled in the trial.

A number of assessments will be conducted before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent form (ICF)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 35-65 years
* Subjects with Omega-3 Index of 5 or less.
* Subjects with Chronic Inflammation Scores of 415 or greater.

Exclusion Criteria:

1. Subjects who are unwilling to provide blood and urine samples during the initial and subsequent test points.
2. Subjects that have consumed Anti-Aging Formula, omega-3 fatty acid (i.e. fish oil, krill oil, algal oil), lutein, zeaxanthin, carotenoids, GLA (borage or evening primrose oils) and/or Vitamin D supplements during the last 3 months
3. Subjects who were ill (i.e. rhino virus, influenza, etc.) within two weeks prior to the study start, or who have any active systemic infection (infected tooth, bladder infection, sinus infection, etc.)
4. Subjects taking:

   1. Anti-inflammatory medications including the nonsteroidal anti-inflammatory drugs (NSAID), cyclooxygenase (COX)-1 and COX-2 inhibitors, such as aspirin, ibuprofen (Advil and Voltaren), and naproxen, and acetaminophen (Tylenol®), either routinely or during the 7 days before baseline urine and blood testing.
   2. H2 antagonist/blockers [e.g. cimetidine (Tagamet®), ranitidine (Zantac®)]
   3. Anti-histamines [e.g. fexofenadine (Allegra®), terfenadine (Seldane®), diphenhydramine (Benadryl®), desloratadine (Clarinex®)], either routinely or during the 7 days before baseline urine and blood testing.
   4. Statins [e.g. atorvastatin (Lipitor®), lovastatin (Altoprev®), pitavastatin (Livalo®), pravastatin (Pravachol®), rosuvastatin (Crestor®), simvastatin (Zocor®)]
   5. Cannabinoids/Cannabis
   6. Corticosteroids including:

      * Inhaled treatments such as beclomethasone (QVAR®), budesonide (Pulmicort®), ciclesonide (Alvesco®), fluticasone (Flovent®), mometasone (Asmanex Twisthaler®)
      * Oral treatments such as Prednisone
      * Injectables such as cortisone injections and IV treatments such as Humira®, Enbrel® and Remicade®
      * Topical treatments such as hydrocortisone (Anusol®)
5. Subjects with known allergy or intolerance to the test material ingredients (i.e. fish, soy)
6. Subjects who consume fish more than twice per week
7. Subjects who smoke tobacco and/or cannabis products
8. Women who are pregnant or are planning to become pregnant or are lactating during the course of the study
9. Subjects who have participated in a clinical trial (CT) within the past 3 months
10. Subjects living in the same household as subjects that are currently enrolled within this study
11. Subjects with diabetes (or taking Metformin), diagnosed arthritis, diagnosed chronic kidney disease, cancer, or with any apparent acute injury inflammation (e.g. torn rotator cuff, broken leg, severe skin abrasions).
12. Subject who consume alcohol during the 12 hours before baseline urine and blood testing

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or Female
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Urinary 1-dehydrothromboxane B2 using The Chronic Inflammation Test | Baseline to 90 days
  The concentration of 1-dehydrothromboxane B2 in urine using The Chronic Inflammation Test (https://chronicinflammationtest.com) after treatment with Anti-Aging Formula, control fish oil and inert placebo.
Omega-3 Index | Baseline to 90 days
  The concentration of EPA+DHA expressed as the Omega-3 index (https://omegaquant.com), after treatment with Anti-Aging Formula, control fish oil and inert placebo
Urinary 8-hydroxy-2' -deoxyguanosine (8- OHdG) | Baseline to 90 days
  The concentration of 8-OHdG in urine after treatment with Anti-Aging Formula, control fish oil and inert placebo.
Urinary 8-isoprostane | Baseline to 90 days
  The concentration of 8-isoprostane in urine after treatment with Anti-Aging Formula, control fish oil and inert placebo.

SECONDARY OUTCOMES:
Blood pressure | Baseline to 90 days
  Blood pressure reported as mmHg (Systolic/Diastolic) after treatment with Anti-Aging Formula, control fish oil and inert placebo.
Resting heart rate | Baseline to 90 days
  Resting heart rate in beats per minute after treatment with Anti-Aging Formula, control fish oil and inert placebo.
Height | Baseline to 90 Days
  Height in meters (m) after treatment with Anti-Aging Formula, control fish oil and inert placebo.
Weight | Baseline to 90 days
  Weight in Kilograms (Kg) after treatment with Anti-Aging Formula, control fish oil and inert placebo.
Body Mass Index (BMI) | Baseline to 90 days
  Weight and height will be combined to calculate BMI as kg/m2 after treatment with Anti-Aging Formula, control fish oil and inert placebo.
General health/function | Baseline to 90 days
  Subjective assessment of general health/function using an in-house designed questionnaire after treatment with Anti-Aging Formula, control fish oil and inert placebo. The questionnaire consists of a list of 27 questions with answers on a scale from 0-4 that cover a variety of health indicators including pain, task oriented performance, mental and emotional well-being, appetite, etc. The resulting score defines General Health/Function as
  * Excellent 81-108
  * Good 54-80
  * Poor 27-53
  * Extremely poor 0-26
Physical activity rating | Baseline to 90 days
  Subjective assessment of physical activity using an in-house designed questionnaire after treatment with Anti-Aging Formula, control fish oil and inert placebo. Results are expressed as how many days per week (0-7) that the Subject exercised to a defined amount, where a greater number of days is considered better.
Perceived health status | Baseline to 90 days
  Subjective assessment of perceived health using an in-house designed questionnaire after treatment with Anti-Aging Formula, control fish oil and inert placebo. The results are expressed as the subjects' perceived health (degrees of good or bad) on the day that the questionnaire is completed using a scale of 0-100 where 0 is the worst imaginable health and 100 is the best imaginable health.
Mental well-being/depression | Baseline to 90 days
  Subjective assessment of mental well-being/depression using the Patient Health Questionnaire-9 after treatment with Anti-Aging Formula, control fish oil and inert placebo. The Patient Health Questionnaire-9 is available in the public domain, and is employed to capture data more focused on mental health indicators of depression. It is a version of the PRIME-MD diagnostic instrument for common mental disorders, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care to monitor severity of depression and response to treatment. Results are presented as a score ranging from 0-27, where 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, and 20-27 is severe depression.
Skin Condition | Baseline to 90 days
  Subjective assessment of skin condition using Observ 520 Skin Analysis (http://www.observ.uk.com/) after treatment with Anti-Aging Formula, control fish oil and inert placebo. Observ 520 Skin Analysis measures skin condition in the epidermal and dermal layers using skin fluorescence and polarized light illumination technology to produce visual indicators of skin's condition.The technology allows overlay of one photo on top of another to enable comparative changes before and after treatment. Numerical data will be created by comparing before and after treatment photos and assigning the descriptors: "improved", "unchanged", or "worsened" that correspond to the values +1, 0, or -1, respectively. The average numerical value from each of the three treatment arms will then be calculated and compared, which will be used as quantitative measures of the treatments' effects on skin condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Connolly, ND, BSc., Principal Investigator — Cornerstone Naturopathic Clinic
Locations (1):
- Cornerstone Naturopathic Clinic, 14 Old School Rd, Upper Tantallon, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morse NL, Reid AJ, St-Onge M. An open-label clinical trial assessing the efficacy and safety of Bend Skincare Anti-Aging Formula on minimal erythema dose in skin. Photodermatol Photoimmunol Photomed. 2018 Mar;34(2):152-161. doi: 10.1111/phpp.12350. Epub 2017 Oct 11. PMID 28884844